CLINICAL TRIAL: NCT02769039
Title: Predictors of Progression to Freezing of Gait in Parkinson's Disease
Brief Title: Predictors of Motor Progression in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1508M77201; 1R01NS088679-01A1 (NIH)
Record Dates: First submitted 2016-04-27; First posted 2016-05-11 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Movement; Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Parkinson's Disease participants: People with early Parkinson's disease with mild-to-moderate severity of disease.
  Interventions: Other: No intervention. Observational studies of sleep, movement and brain imaging
- Control participants: Volunteers who are age (+/- 3 years) and sex matched to the participants with Parkinson's disease
  Interventions: Other: No intervention. Observational studies of sleep, movement and brain imaging

INTERVENTIONS:
Other: No intervention. Observational studies of sleep, movement and brain imaging — Participants will be asked to visit the University for 3 baseline visits which include a screening visit & sleep study, movement tests and magnetic resonance imaging (MRI) scans. Three years later the participant will be asked to repeat the same visits.

SUMMARY:
Treatment resistant motor features, such as postural instability and freezing of gait are common in people with Parkinson's disease and major contributors to morbidity and mortality. This project will use sleep studies, quantitative motor assessments and magnetic resonance imaging to examine the relationship between abnormally increased muscle activity during rapid eye movement sleep and the development and progression of treatment-resistant postural instability and gait disturbances. Specifically, the investigators will test the hypothesis that anticipatory postural adjustments (weight and pressure shifts) during gait initiation are significantly reduced in people with Parkinson's disease who have abnormally elevated muscle activity during rapid eye movement (REM) sleep compared to individuals will Parkinson's disease whose REM sleep muscle activity is normal. In addition, the investigators will test the hypothesis that the level of RSWA at baseline is predictive of measures of motor decline (postural stability and gait) and alterations in the structure and function of locomotor brainstem networks. Since sleep disorders can emerge years before a diagnosis of Parkinson's disease, establishment of a link between sleep and treatment-resistant posture and gait disorders will help identify individuals at risk of developing these disabling motor features of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's Disease (PD).
2. Age 21-75 years
3. Able to ambulate independently without the use of an assistive device (e.g. cane)

Exclusion Criteria:

1. History of Dementia
2. History of musculoskeletal disorders that adversely affects walking and/or balance
3. Other significant neurological disorders
4. Implanted deep brain stimulator(s) (DBS) or other neurosurgeries to treat PD
5. MRI exclusion for 7 tesla scans: presence of any metallic clips or implantable medical devices
6. Pregnant women

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Magnitude of the center of pressure shift during gait initiation. | Measured at baseline (time 0).
  The magnitude of the center of pressure shift during gait initiation is calculated as the displacement of the center of pressure signal from quiet standing (baseline) to the peak lateral and posterior excursion during the anticipatory postural adjustment phase of gait initiation.
Correlation between measures of REM sleep without atonia (RSWA) at baseline and change in the magnitude of the center of pressure shift during gait initiation over the course of 3 years. | Change in magnitude over the course of 3 years
  A linear correlation analysis will be conducted between measures of RSWA at baseline versus the change in shift of the center of pressure during gait initiation between baseline and year 3.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided